CLINICAL TRIAL: NCT01405716
Title: Effectiveness of a Mind-Body Program for Older Adults With Chronic Low Back Pain
Brief Title: Aging Successfully With Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Natalia Morone, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO09100150; R01AG034078-01 (NIH)
Record Dates: First submitted 2011-07-25; First posted 2011-07-29 (Estimated); Last update posted 2017-10-03 (Actual); Status verified 2017-09

CONDITIONS: Low Back Pain
Keywords: Mindfulness; Back Pain; Older adults
MeSH Terms: conditions — Low Back Pain; Back Pain | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Behavioral-Mindfulness (Active Comparator): Mindfulness Meditation
  Interventions: Behavioral: Mindfulness Meditation
- Behavioral-Health (Placebo Comparator): Health Education Class
  Interventions: Behavioral: Health Education

INTERVENTIONS:
Behavioral: Mindfulness Meditation — 8-week mindfulness based program will be compared to and education control group
  Arms: Behavioral-Mindfulness
Behavioral: Health Education — 8-week health education program
  Arms: Behavioral-Health

SUMMARY:
The primary objective of this study is to determine the effectiveness of a mind-body program in increasing function and reducing pain among older adults with chronic low back pain

DETAILED DESCRIPTION:
Among mind-body therapies, there is evidence for an association between pain reduction and mindfulness meditation. Mindfulness meditation provides a potentially safe, effective, nonpharmacologic, noninvasive, simple method for pain relief and increased function that could be used for the frailest older adult. This experimental study is designed as a randomized, education controlled clinical trial of a mind-body program for older adults with chronic low back pain. A sample of 300 independent, community-dwelling adults 65 years of age and older will be recruited. After determining eligibility, study participants will give written informed consent and will be randomized to either the mindfulness-based stress reduction (MBSR) program or the health education control program. Participants in the mind-body group will receive the intervention of eight weekly 90-minute mindfulness meditation sessions that are modeled on the MBSR program. Controls will receive an 8-week health education program based on the 10 Keys(TM) to Healthy Aging. After completion of the 8-week program, participants in both programs will be asked to return for 12 monthly booster sessions. Prior to initiating the program, immediately after the last program session, and 6 & 12 months later, the following parameters will be assessed: (1) physical function, (2) pain severity, (3) neuropsychological performance, (4) measures of mindfulness, (5) demographic factors, and (6) biomedical factors.

ELIGIBILITY:
Inclusion Criteria:

* 65 years or older
* Have intact cognition (Mini-Mental Status Exam (MMSE) >24)
* 65 years of age or older.
* Have functional limitations due to their low back, defined as a score of at least 12 on the Roland and Morris Disability Questionnaire.
* CLBP, defined as moderate pain occurring daily or almost every day for at least the previous three months.
* Speak English.

Exclusion Criteria:

* Do not meet the above inclusion criteria
* Have previously participated in a mindfulness meditation program.
* Have serious underlying illness (like malignancy, infection, unexplained fever, weight loss or recent trauma) causing their pain.
* Are non-ambulatory, or have severely impaired mobility (i.e., require the use of a walker): since measurement of physical performance in the proposed study includes timed chair rise, gait velocity, and standing balance, conditions other than back pain that could negatively impact these measures may confound our study results.
* Have severe visual or hearing impairment: since this study will involve questionnaires and telephone evaluations, severe visual and/or hearing impairments may interfere with data collection and data validity. For example, the Mini-Mental Status Exam has never been validated in those with severe visual or hearing disturbance.
* Have pain in other parts of the body that is more severe than their low back pain, [defined as pain other than in the lower back that occurs daily or almost every day and is of at least moderate intensity] or acute back pain: since we will be specifically evaluating chronic low back pain, we do not want to confound the outcome data with [significant pain] from other areas or with acute pain. Thus only participants with chronic low back pain severity that is greater than pain severity elsewhere in the body will be included.
* Have acute or terminal illness: To insure weekly participation and a twelve month follow-up, participants with an acute or terminal illness will be excluded from the study.
* Have moderate to severe depression, defined as a Geriatric Depression Scale score of 21 and above: since active depression may affect the psychological outcomes of the study and may affect compliance with participation in the intervention and control programs.
* Do not have access to a telephone: since monthly assessments will be done over the telephone.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 282 (Actual)
Dates: Start 2011-02; Primary Completion 2014-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change in the Roland-Morris Questionnaire | Change from Baseline to 8-weeks to 6-months to 12-months
  The Roland-Morris Questionnaire is a disability measure in which greater levels of disability are reflected by higher numbers on a 24-point scale. The RMQ has been shown to yield reliable measurements, which are valid for inferring the level of disability, and to be sensitive to change over time for groups of patients with low back pain

CONTACTS AND LOCATIONS:
Overall Officials: Dr Natalia Morone, MD, MS, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Morone NE, Greco CM, Moore CG, Rollman BL, Lane B, Morrow LA, Glynn NW, Weiner DK. A Mind-Body Program for Older Adults With Chronic Low Back Pain: A Randomized Clinical Trial. JAMA Intern Med. 2016 Mar;176(3):329-37. doi: 10.1001/jamainternmed.2015.8033. PMID 26903081
- [Derived] Morone NE, Greco CM, Rollman BL, Moore CG, Lane B, Morrow L, Glynn NW, Delaney J, Albert SM, Weiner DK. The design and methods of the aging successfully with pain study. Contemp Clin Trials. 2012 Mar;33(2):417-25. doi: 10.1016/j.cct.2011.11.012. Epub 2011 Nov 15. PMID 22115971